CLINICAL TRIAL: NCT07206537
Title: The Role of Vitamin K2 in Preventing Glucocorticoid-Induced Bone Loss in Children With Nephrotic Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FMASU MD189/2025
Record Dates: First submitted 2025-09-26; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Pediatrics Nephrology
Keywords: Nephrotic Syndrome; Vitamin K2
MeSH Terms: conditions — Nephrotic Syndrome | interventions — Vitamin K 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): 30 Nephrotic patients of matched age and sex of the cases have been on Glucocorticoids for 6 months or more not receiving vitamin k2 supplements
- Case (Active Comparator): 30 Nephrotic patients of matched age and gender who have been on Glucocorticoids for 6 months or more, receiving vitamin k2 supplements for 24 weeks.
  Interventions: Drug: Vitamin K 2

INTERVENTIONS:
Drug: Vitamin K 2 — Oral vitamin K2 supplementation
  Arms: Case

SUMMARY:
Long-term glucocorticoids therapy is associated with various complications, including decreased bone strength (Glucocorticoid-induced osteoporosis) and an increased risk of fracture.

Vitamin K2 has been recently deemed appreciable as a topic of research as it plays a pivotal role in maintenance of the bone strength, and it has been proved to have a positive impact on the bone metabolism.

This study examines the impact of oral vitamin K2 supplementation on bone metabolism in pediatric patients with nephrotic syndrome on long-term steroid therapy, offering valuable therapeutic insights

DETAILED DESCRIPTION:
Nephrotic syndrome is the predominant glomerular disorder in pediatric patients. It is defined as nephrotic-range proteinuria and either hypoalbuminemia (serum albumin <30 g/l (3 g/di)) or edema when albumin level is not available. Nephrotic-range proteinuria is defined as first morning urine or *24-h urine protein-creatinine ratio (uPCR) ≥ 2g/g (or 200 mg/mmol or ≥ 3+ dipstick).

Steroids are the first-line treatment for nephrotic syndrome, with an initial regimen of daily prednisolone/prednisone at a dose of 60 mg/m2/day for at least 4 weeks followed by an alternate-day regimen for several weeks. While effective in managing symptoms, glucocorticoids directly inhibit bone formation by decreasing osteoblast differentiation and by inhibition of type 1 collagen synthesis. It also stimulates bone resorption by directly enhancing osteoclast activity, as well as indirectly via increased PTH production and decreased gonadotropins, resulting in glucocorticoid-induced osteoporosis (GIOP).

In pediatric patients, the growing skeleton is especially vulnerable to these effects, and early intervention is crucial to prevent long-term complications, a clinical study reported increased fracture risk in children who require more than four courses of GCs. In general, bone loss caused by GC treatment occurs within the first 6 months of treatment.

Vitamin K, a lipid-soluble vitamin, is an essential micronutrient. It includes:

* Vitamin K1 (phylloquinone): Found primarily in green leafy vegetables.
* Vitamin K2 (menaquinones, MKs): Includes 13 types, found in meat, fermented food and cheese and predominantly produced by colonic bacteria, except for MK-4, which is synthesized in animal tissues through tissue-specific conversion of vitamin K1.
* Vitamin K3 (menadione): A synthetic form of the vitamin. Among the menaquinones, MK-7 is the most active form due to its superior absorption (peaking at 4 hours), longer half-life (72 hours) and better bioavailability. Additionally, MK-7 has fewer side effects compared to other forms.

In this context, Vitamin K2 promotes bone formation by stimulating the osteoblasts differentiation, increasing the level of some bone formation markers (e.g., alkaline phosphatase and insulin-like growth factor), and regulating the extracellular matrix mineralization through Y-glutamyl carboxylation. Additionally, vitamin K prevents bone resorption via its anticatabolic activities, namely, decreasing osteoclasts differentiation and inhibiting osteoblasts apoptosis.

So vitamin K2 supplementation may serve as a multifaceted intervention in managing the long-term side effects of glucocorticoid therapy in pediatric nephrotic syndrome patients.

Alkaline phosphatase is a glycoprotein that is connected to the surface of cells. In humans ALP is expressed in four gene loci code: nonspecific, intestinal, placental and germ cells. Nonspecific gene is synthesized in a variety of tissues (bone, kidney, liver and early placenta) . Bone specific alkaline phosphatase (BALP) has been used due to its high sensitivity as a bone formation marker. It is produced by osteoblasts and is involved in the calcification of bone matrix. It has been reported that low BALP level had a sensitivity of 100%, a specificity of 94% and a positive predictive value of 72% in the prediction of low-turnover bone disease.

Tartrate-resistant alkaline phosphatase (TRAP) is a glycoprotein produced by mature osteoclasts, activated dendritic cells, and macrophages, therefore TRAP is an indicator of osteoclast and macrophage activity. There are two known isoforms (TRAP5a,b). TRAP5b is a specific biomarker of osteoclastic resorption activity, while TRAP5a is a non-osteoclastic form.

ELIGIBILITY:
Inclusion Criteria:

* Nephrotic patients under 16 years of age of both genders who were treated with GC for the first time. GC treatment was initiated at a dose of 2 mg/kg/day prednisolone with gradual dose reduction.
* All patients have been on glucocorticoid therapy for more than 6 months. All patients have sufficient vitamin D level 30 ng/ml (75 nmol/L) or above.

Exclusion Criteria:

1. Patients with impaired kidney functions.
2. Non-compliant patients on medications or vitamin supplements.
3. Diseases that affect fat-soluable vitamins absorption such as gallbladder or biliary disease, cystic fibrosis, celiac disease, etc.
4. History of vitamin K-related disorders as bleeding disorders, osteomalacia , etc.
5. History of bone fracture before the study.
6. Any nephrotic syndrome with identified genetic causes.

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Prevention of Glucocorticoid-Induced Bone Loss | 6 month
  To assess the impact of vitamin K2 supplementation on glucocorticoid-induced bone loss in pediatric patients with nephrotic syndrome.
  To determine the effect of vitamin K2 on specific biochemical markers of bone turnover (e.g., bone-specific alkaline phosphatase , tartrate-resistant acid phosphate) in the study population

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt